CLINICAL TRIAL: NCT02223949
Title: Labor Induction and Maternal BMI: Comparison of Different Pre-induction Cervical Ripening Methods: The Cook Double Balloon Catheter vs PGE1 Tablets in Lean, Overweight, and Obese Women. A Prospective Randomized Study.
Brief Title: Labor Induction and Maternal BMI, Comparison of Different Pre-induction Cervical Ripening Methods
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0033-14-HYMC
Record Dates: First submitted 2014-08-21; First posted 2014-08-22 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Obesity; Labor Complications
Keywords: Obesity; Labor complications; Induction of labor; Mechanical cervical ripening
MeSH Terms: conditions — Obesity; Obstetric Labor Complications | interventions — Alprostadil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cook double balloon catheter (Experimental): Insertion of the Cook double balloon catheter to the cervix until both balloons are properly located in the cervical canal. After properly located it is inflated with 20 ml of saline. Then both balloons are additionally inflated to a total of 80 ml each balloon. Twelve hours later the balloons are deflated and the device is removed.
  Interventions: Device: Cook double balloon catheter
- PGE1 tablet insertion (Active Comparator): Insertion of 25 mg PGE1 (Prostaglandin E1) tablet is inserted in the posterior fornix. The patient woll the be instructed to stay in bed for the next 60 minutes. After six hours a repeated dose will be administered. Total of 4 PGE1 doses within 24 hours.
  Interventions: Drug: PGE1 tablet

INTERVENTIONS:
Device: Cook double balloon catheter
  Arms: Cook double balloon catheter
Drug: PGE1 tablet
  Other Names: Prostaglandin E1
  Arms: PGE1 tablet insertion

SUMMARY:
The purpose of this study is to investigate whether mechanical cervical ripening (using the Cook double balloon catheter) is superior or inferior to pharmacological agents (PGE1) in overweight and obese women undergoing labor induction.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years of age or older.
* Diagnosed to be pregnant (al least 37 weeks of gestation) with a medical indication for labor induction, including: postdate pregnancy, preeclampsia, gestational or chronic hypertension, Gestational Diabetes Mellitus at term, Oligohydramnios, Polyhydramnios, fetal growth restriction, maternal background disease necessitating delivery, Isoimmunisation, maternal Thrombophilia, intrahepatic cholestasis of pregnancy.
* Having a Bishop score of 4 points or less.
* Diagnosed as having singleton pregnancy at term (37 weeks at least) in a vertex presentation, with intact membranes, and absence of significant regular uterine contraction.
* Willingness to comply with the protocol for the duration of the study.
* Has agreed and signed an informed consent after given oral and written explanation.

Exclusion Criteria:

* Anay contraindication for a vaginal delivery (i.e. placenta previa, non vertex presentation, estimated fetal weight of less than 4500 gr).
* Ruptured membranes.
* Previous cesarian section or presence of any uterine scar.
* Documented labor with four or more spontanous uterine contractions per hour.
* Suspected fetal distress necessitating immediate intervention.
* Proven malignancy of the cervix.
* Active vaginal bleeding.
* Active inflammatory or purulent condition of the lower genital tract.
* Active asthma.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 624 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-10 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Cesarian section rate | 24 hours

SECONDARY OUTCOMES:
Incidence of excessive uterine activity Incidence of excessive uterine activity | 24 hours
  At least 6 uterine contractions per 10- minutes period, or hyperstimulation, if combined with fetal heart rate abnormalities, or hypertonus defined as single contraction of 2-minute duration.
Active labor onset | 24 hours
Proportion of vaginal delivery | 24 hours
Treatment failure | 12-24 hours
  Proportion of subjects with unfavorable/unchanged Bishop score 12-24 hours after ripening
The ripening-to-delivery time interval | 24 hours
Need for oxytocin induction and/or augmentation of labor | 24 hours
Mode of delivery | 24 hours
  NVD vs. instrumental
Intra-partum or postpartum fever | 48 hours
Incidence of meconium staining | 24 hours
The proportion of neonates with 5-minute Apgar scores of less than 7 | 48 hours
The number of neonates who were admitted to the neonatal intensive care unit | 48 hours
morbidity and mortality | 48 hours
  Number of cases of serious maternal and/or neonatal morbidity or death (including uterine rupture, maternal admission to the intensive care unit, maternal septicemia, placental abruption, hemorrhage at required blood transfusion, hysterectomy, neonatal seizures, birth asphyxia, meconium aspiration syndrome, or neonatal sepsis).

CONTACTS AND LOCATIONS:
Overall Officials: Saja Murra Anabosy, MD, Principal Investigator — Hillel Yaffe Medical Center; Asnat Walfisch, MD, Study Chair — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel

REFERENCES:
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264